CLINICAL TRIAL: NCT04707729
Title: ROX Index Compared to Standard of Care for the Timing of Intubation in Patients Supported by Nasal High Flow: a Randomized Controlled Trial
Brief Title: ROX Index for the Timing of Intubation in Nasal High Flow
Acronym: ROX-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AG)454/2020
Record Dates: First submitted 2020-12-24; First posted 2021-01-13 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Acute Hypoxemic Respiratory Failure
Keywords: High flow nasal cannula; Nasal high flow; High flow oxygen therapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: The ROX-1 trial is an international, multicenter, parallel, open-label randomized controlled two-arm trial that will be performed in patients with AHRF, supported by nasal high flow, who are admitted to the intensive care unit (ICU).
  Patients will be randomized after stratification according to PaO2/FiO2, through an online automatic centralized and computerized system to one of the study groups (1:1 ratio): traditional intubation criteria or traditional intubation criteria + ROX criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients will be intubated according to both the standard of care
- Standard of care + ROX algorithm (Experimental): In the intervention arm, patients will be intubated according to both the standard of care and the ROX index, whichever are met first. If the patient has a ROX index below different thresholds after different time-point within the first 12 hours since randomization, the NHF support will be increased to the maximum tolerated flow (up to 60L/min) and FIO2 of 1 and subsequently titrated with the target SpO2. Then, the ROX index will be recalculated in 30 minutes. If the patient is already treated with to 60L/min) and FIO2 of 1 and no further increase could be done, the ROX index will be recalculated after 30 minutes of full NHF support. Then: 1) if the ΔROX is <0 the patient will be intubated; 2) if the ΔROX is 0-0.5, the ΔROX will be reassessed in 30 minutes; and 3) if the ΔROX is >0.5 the patient will not be intubated, NHF will be managed as protocolized and respiratory condition will be reassessed every two hours or at any new clinical deterioration.
  Interventions: Diagnostic Test: ROX index algorithm

INTERVENTIONS:
Diagnostic Test: ROX index algorithm — The thresholds of the ROX index for intubation are the following:
  * After 2 hours of HFNC: ROX <2.85.
  * After 4 and 6 hours of HFNC: ROX <3.47
  * After 8, 10 and 12 hours of HFNC: ROX <3.85 If the ROX index is between the abovementioned thresholds and 4.88, the NHF support will be also increased to the maximum tolerated flow (up to 60L/min) and FIO2 of 1 and subsequently titrated with the target SpO2. If the patient is already treated with to 60L/min) and FIO2 of 1 and no further increase could be done and the ROX index will be recalculated after 30 minutes of full NHF support. The ROX index will be recalculated in 30 minutes: 1) if the ΔROX is <0 the patient will be intubated; 2) if the ΔROX is 0-0.5, the ΔROX will be reassessed in 20 minutes; and 3) if the ΔROX is >0.5 the patient will not be intubated, NHF will be managed as protocolized and respiratory condition will be reassessed every two hours or at any new clinical deterioration.
  Arms: Standard of care + ROX algorithm

SUMMARY:
Late or delayed intubation in patients with acute hypoxemic respiratory failure (AHRF) treated with nasal high flow (NHF) is associated with increased patient mortality. The ROX index has been designed and validated to predict outcome of NFH therapy by identifying those patients with a high risk of NHF failure and those with a high probability of success. Whether or not the ROX index may improve patient outcome remains to be shown. To do so, a strategy using the ROX index must lead to earlier intubation than commonly-used criteria.

The objective of the ROX-1 trial is to assess whether the use of an algorithm incorporating the ROX index to standard of care for the time to intubation in patients with AHRF supported with NHF isassociated with an increase in the proportion of patients who are intubated within the first 12 hours among those patients who fail on NHF.

DETAILED DESCRIPTION:
This is a pilot study to assess whether the use of an algorithm incorporating the ROX index to traditional criteria for intubation in patients with AHRF supported with NHF is:(i) feasible; (ii) associated with a decreased time to intubation.

The ROX-1 trial is an international, multicenter, parallel, open-label randomized controlled two-arm trial that will be performed in patients with AHRF, supported by nasal high flow, who are admitted to the intensive care unit (ICU). Ethics approval will be sought from each participating institution before starting enrolmentand consent will be obtained for each patient. The coordinating center will be Hospital Universitari Vall d'Hebron in Barcelona, Spain.

All consecutive patients older than 18 years with acute hypoxemic respiratory failure who need to be supported with nasal high flow (NHF) will be enrolled if they meet all the following criteria:

1. Respiratory rate > 25 breaths/min
2. A pulse oximetry (SpO2)<92% while receiving standard oxygen administered through a facemask at 10L/min or more.
3. Pulmonary infiltrate on chest X-ray.

Patients already treated with NHF for acute respiratory failure prior to ICU admission will be enrolled if duration of NHF prior to randomization does not exceed one hour.

Non-inclusion criteria are: Patients younger than 18 years old, Patients with indication for immediate intubation, patients with do not intubate order, patients electively intubated for diagnostic or therapeutic procedure (fibrobronchoscopy, surgery), patient with post-extubation AHRF, awake ECMO, pregnancy and refusal to participate or participation in another interventional study with the same primary outcome. Reasons for non-inclusion in screend patients will be registered.

Patients admitted to the ICU with acute hypoxemic respiratory failure will be screened, included after having received study information, and signed informed consent. They will be randomized after stratification according to PaO2/FiO2, through an online 4 automatic centralized and computerized system to one of the study groups (1:1 ratio): traditional intubation criteria or traditional intubation criteria + ROX criteria. Due to the nature of the intervention, blinding will not be feasible.

Randomization will be stratified to PaO2/FiO2 in order to analyse separately those patients with a PaO2/FiO2 ratio ≤ 200 and > 200. Intubation criteria for each study arm HFNC failure will be defined as the subsequent need for invasive MV. After randomization, clinicians will set NHF to the maximum tolerated flow (up to 60L/min) and FIO2 will be titrated targeting a SpO2 between 94-98% (88-92% in case of underlying chronic lung disease). In both groups, the presence of intubation criteria will be assessed every two hours during the first 12 hours after randomization and after any clinical deterioration. Between 12 and 24 hours of NHF therapy, the presence of intubation criteria will be assessed every 4 hours. Beyond the first 24 hours after randomization, the presence of intubation criteria will be assessed once a day and after any clinical deterioration.

In the intervention arm, patients will be intubated according to both the traditional intubation criteria and the ROX index, which ever are met first. Moreover, during the first two hours of NHF supportive therapy after randomization, the ROX index will be measured every 30 minutes. If the patient has a ROX index <2.85, the NHF support will be increased to the maximum tolerated flow (up to 60L/min) and FIO2 of 1 and subsequently titrated with the target SpO2. Then, the ROX index will be recalculated in 30 minutes. If the patient is already treated with to 60L/min and FIO2 of 1 and no further increase could be done, the ROX index will be recalculated after 30 minutes of full NHF support. Then: 1) if the ΔROX is <0 the patient will be intubated; 2) if the ΔROX is 0-0.5, the ΔROX will be assessed in 30 minutes; and 3) if the ΔROX is >0.5 the patient will not be intubated, NHF will be managed as protocolized and respiratory condition will be reassessed every two hours or at any new clinical deterioration.

Between the 2 and 6 hours after randomization, the ROX index will be measured every 60 minutes. If the ROX index is <3.47, the NHF support will be also increased to the maximum tolerated flow (up to 60L/min) and FIO2 of 1 and subsequently titrated with the target SpO2. If the patient is already treated with to 60L/min and FIO2 of 1 and no further increase could be done and the ROX index will be recalculated after 30 minutes of full NHF support. As described before, the ROX index will be recalculated in 30 minutes: 1) if the ΔROX is <0 the patient will be intubated; 2) if the ΔROX is 0-0.5, the ΔROX will be reassessed in 20 minutes; and 3) if the ΔROX is >0.5 the patient will not be intubated, NHF will be managed as protocolized and respiratory condition will be reassessed hourly or at any new clinical deterioration.

Finally, between the 6 and 12 hours after randomization, the ROX index will be measured every 60 minutes. If the ROX index is <3.85, the NHF support will be increased to the maximum tolerated flow (up to 60L/min) and FIO2 of 1 and subsequently titrated with the target SpO2. If the patient is already treated with to 60L/min) and FIO2 of 1 and no further increase could be done and the ROX index will be recalculated after 30 minutes of full NHF support. Then, the ROX index will be calculated in 30 minutes and decision of intubation will be taken according to the previously described ΔROX. In the ROX group, if there is any clinical deterioration beyond the first 12 hours of treatment , the algorithm should be restarted from the beginning, considering time 0 as the time when new clinical deterioration started. End of follow-up. Enrolled patients will be followed for one month or until ICU discharge or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients older than 18 years with acute hypoxemic respiratory failure who need to be supported with nasal high flow (NHF) will be considered for inclusion.

  * Criteria for initiation of NHF if they had a respiratory rate > 25 breaths/min and/or pulse oximetry (SpO2) < 92% while receiving standard oxygen administered through a facemask at 10 L/mn or more.
  * Patients already treated with NHF for acute respiratory failure prior to ICU admission will be enrolled if duration of NHF prior to randomization does not exceed one hour.

Exclusion Criteria:

* Patients younger than 18 years old.
* Patients with indication for immediate intubation.
* Patients treated with NHF for more than 1h prior to randomization.
* Patients with do-not-intubate order.
* Patients electively intubated for diagnostic or therapeutic procedures. (fibrobronchoscopy, surgery).
* Patients with no pulmonary infiltrates on chest X-ray
* Patient with post-extubation AHRF.
* Awake ECMO.
* Pregnancy.
* Refusal to participate or participation in another interventional study with the same primary outcome.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Early intubation | 12 hours since HFNC onset
  Proportion of patients who will be intubated in the first 12 hours after inclusion between the two groups

SECONDARY OUTCOMES:
Intubation rate | Through ICU length of stay, an average of 30 days
  Rate of total intubations (early plus late)
28-day mortality | 28 days
  Mortality within the first 28 days since randomization
90-day mortality | 90 days
  Mortality within the first 90 days since randomization
ICU mortality | Through ICU length of stay, an average of 30 days
  Mortality in the ICU
Hospital mortality | Through hospital length of stay, an average of 45 days
  Mortality in the hospital
Ventilator-free days within the first 28 days | 28 days since the intubation
  Days free of mechanical ventilation in the first 28 days in those patients who needed to be intubated
Days free of respiratory support within the first 28 days | 28 days since randomization
  Days free of respiratory support (including HFNC, CPAP, NIV or invasive mechanical ventilation) in the first 28 days
Use of rescue treatments | Through ICU length of stay, an average of 30 days
  Need for rescue therapies for refractory hypoxemia
Need for tracheotomy | Through ICU length of stay, an average of 30 days
  Need for tracheotomy
ICU length of stay | Through ICU length of stay, an average of 30 days
  Days admitted in the ICU
Hospital length of stay | Through hospital length of stay, an average of 45 days
  Days admitted in the hospital
Rate of complications during tracheal intubation | Through ICU length of stay, an average of 30 days
  Proportion of complications that appear during endotracheal intubation in those patients who fail

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Roca, MD PhD, Principal Investigator — Universitat Autònoma de Barcelona (UAB)
Locations (12):
- Rush University Chicago Hospital, Chicago, Illinois, United States
- China (3):
  - First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Second Military Medical University Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
- Spain (8):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de Ciudad Real, Ciudad Real
  - Hospital Civil Fray Antonio Alcalde, Guadalajara
  - Hospital Son Llàtzer, Palma de Mallorca
  - Hospital Parc Taulí, Sabadell
  - Hospital Moisès Broggi, Sant Joan Despí
  - Hospital Virgen de la Salud, Toledo

REFERENCES:
- [Background] Brochard L, Mancebo J, Wysocki M, Lofaso F, Conti G, Rauss A, Simonneau G, Benito S, Gasparetto A, Lemaire F, et al. Noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 1995 Sep 28;333(13):817-22. doi: 10.1056/NEJM199509283331301. PMID 7651472
- [Background] Roca O, Caralt B, Messika J, Samper M, Sztrymf B, Hernandez G, Garcia-de-Acilu M, Frat JP, Masclans JR, Ricard JD. An Index Combining Respiratory Rate and Oxygenation to Predict Outcome of Nasal High-Flow Therapy. Am J Respir Crit Care Med. 2019 Jun 1;199(11):1368-1376. doi: 10.1164/rccm.201803-0589OC. PMID 30576221
- [Background] Roca O, Messika J, Caralt B, Garcia-de-Acilu M, Sztrymf B, Ricard JD, Masclans JR. Predicting success of high-flow nasal cannula in pneumonia patients with hypoxemic respiratory failure: The utility of the ROX index. J Crit Care. 2016 Oct;35:200-5. doi: 10.1016/j.jcrc.2016.05.022. Epub 2016 May 31. PMID 27481760